CLINICAL TRIAL: NCT05978089
Title: Efficacy and Safety of Yangxinshi Tablet in Improving Exercise Tolerance in Patients With Chronic Coronary Syndrome(Qi Deficiency and Blood Stasis Syndrome):A Randomized, Double-blind,Placebo-parallel-controlled,Multicenter Clinical Study
Brief Title: Effect of Yangxinshi Tablet on Exercise Tolerance in Patients With Chronic Coronary Syndrome（MET STUDY）
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Wang Xian, Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Growful2201YXS
Record Dates: First submitted 2023-07-16; First posted 2023-08-07 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Chronic Coronary Syndrome
Keywords: Cardiopulmonary Exercise Test; Yangxinshi
MeSH Terms: interventions — Yangxinshi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Yangxinshi tablets
  Interventions: Drug: Yangxinshi tablet
- Control group (Placebo Comparator): Yangxinshi tablet simulants
  Interventions: Drug: Yangxinshi tablet simulants

INTERVENTIONS:
Drug: Yangxinshi tablet — The treatment group was given Yangxinshi tablets (3 tablets/time and 3 times/day). The treatment period was 24 weeks.
  Other Names: Yangxinshi
  Arms: Treatment group
Drug: Yangxinshi tablet simulants — The control group was given Yangxinshi tablet simulants (3 tablets/time and 3 times/day).The treatment period was 24 weeks.
  Arms: Control group

SUMMARY:
This study adopted a randomized, double-blind, placebo-controlled, multicenter clinical design and compared the effects of Yangxinshi tablet and placebo on exercise tolerance in patients with chronic coronary syndrome (CCS).

DETAILED DESCRIPTION:
The aim of the research is to find out if the addition of Yangxinshi tablets on the basis of conventional treatment can improve exercise tolerance of patients with chronic coronary syndrome (CCS), improve quality of life and mental health. A total of 120 qualified CCS patients were randomly divided into two groups. In addition to conventional treatment, the experimental group was given Yangxinshi tablets (3 tablets/time and 3 times/day), and the control group was given Yangxinshi tablet simulants (3 tablets/time and 3 times/day). The treatment period was 24 weeks. The primary endpoints were metabolic equivalents (METs), and peak oxygen uptake measured by cardiopulmonary exercise testing after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria must be met to participate in the study:

1. Meet the diagnostic criteria for CCS in Western medicine; stable coronary heart disease (CHD) with a degree of coronary stenosis ≥50% by angiography or computed tomography angiography (CTA) (including patients with more than 1 year of revascularization)
2. Meet the TCM standard of Qi deficiency and blood stasis syndrome
3. MET < 5 measured by cardiopulmonary exercise test (treadmill)
4. Age between 18 and 75 years (including both age limits), with no limitation on sex
5. Understanding and voluntarily signing the written informed consent

Exclusion Criteria:

All the following criteria must not be met to participate in the study:

1. Individuals with lower extremity dysfunction, intermittent claudication or severe leg pain who cannot participate in cardiopulmonary exercise tests
2. Individuals with acute coronary syndrome within 1 month after percutaneous coronary intervention (PCI) or within 3 months after coronary artery bypass grafting (CABG)
3. Individuals with serious primary diseases related to the liver, kidney, and hematopoietic system, acute infectious diseases, and mental illness and individuals with other diseases who are not suitable for cardiopulmonary exercise tests
4. Individuals with a revascularization plan within a month
5. Individuals with left main stenosis ≥50% or proximal left anterior descending (LAD) diameter stenosis ≥90% without PCI or CABG
6. Individuals with absolute and relative contraindications to cardiopulmonary exercise testing (please see Appendix 11 for details)
7. Individuals with New York Heart Association (NYHA) cardiac function class III and IV
8. Individuals with acute cerebrovascular disease
9. Individuals with uncontrolled hypertension: systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 100 mmHg
10. Individuals found to be in a state of severe anxiety and depression as determined using the GAD-7 and PHQ-9
11. Individuals with allergies or abnormal drug reactions to the test drugs
12. Women of childbearing age who are pregnant or breastfeeding, plan to get pregnant within six months, have a positive pregnancy test, and cannot take effective contraceptive measures during the study period
13. Individuals who have regularly taken YTs, Chinese herbal decoctions or proprietary Chinese medicines with similar curative effects within the past 7 days (please refer to Appendix 12 for the names of proprietary Chinese medicines)
14. Individuals who have participated in other clinical trials within the past 3 months
15. Individuals unsuitable for the clinical trials, as determined by the researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test (treadmill): (MET and peak oxygen uptake) | 24 weeks
  MET=Metabolic Equivalent of Task

SECONDARY OUTCOMES:
anaerobic threshold | 24 weeks
  Cardiopulmonary exercise test (treadmill)
oxygen pulse | 24 weeks
  Cardiopulmonary exercise test (treadmill)
maximal exercise ventilation | 24 weeks
  Cardiopulmonary exercise test (treadmill)
electrocardiogram (ECG) | 24 weeks
  Start time and duration determined by 1-mm downward shift in the ST segment on the electrocardiogram (ECG) during the cardiopulmonary exercise test
CCS angina classification | 24 weeks
  The change in Canadian Cardiovascular Society (CCS) angina scores in all participants. Scoring is via Class I-IV where class IV is worse outcome.
Seattle Angina Questionnaire | 24 weeks
  The Seattle Angina Questionaire (SAQ) quantifies patients'physical limitations caused by angina. The scale is transformed to a score of 0 to 100, where higher scores indicate better function (less physical limitation)
Pittsburgh Sleep Quality Index (PSQI) | 24 weeks
  score range: 0~21，higher scores mean a worse outcome.
General Anxiety Disorder-7 (GAD-7) | 24 weeks
  score range: 0~21，higher scores mean a worse outcome.
Patient Health Questionnaire (PHQ-9) | 24 weeks
  score range: 0-27，higher scores mean a worse outcome.
Traditional Chinese medicine (TCM) Syndrome Score | 24 weeks
  the main symptoms score range: 2-6，the secondary symptoms score range: 1-3，higher scores mean a worse outcome.
Hospitalization within 6 months of taking the medicine | 24 weeks
  total hospitalization time and hospitalization frequency

OTHER OUTCOMES:
Liver function | 24 weeks
  alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), total bilirubin (TBil), and glutamyl transferase (GGT) (γ-GT)
Renal function | 24 weeks
  blood urea nitrogen (BUN) and serum creatinine (Scr)
Myocardial markers | 24 weeks
  creatine kinase (CK), troponin I (TnI) (if not available, troponin T (TnT)), and N-terminal pro-B-type natriuretic peptide (NT-proBNP)
Blood lipids | 24 weeks
  cholesterol (CHO), triglyceride (TG), high-density lipoprotein (HDL), and low-density lipoprotein (LDL)

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xian, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (6):
- China (6):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Dongzhimen Hospital Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of CM, Zhengzhou, Henan